CLINICAL TRIAL: NCT00939705
Title: Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Topiramate (2 x 25 mg), Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Topamax®, Ortho-McNeil Neurologics, Inc.) in Fed, Healthy, Adult Subjects
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Ltd.'s Topiramate Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 06TOR02
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
MeSH Terms: interventions — Topiramate

ARMS (2):
- Torrent Topiramate (Experimental)
  Interventions: Drug: topiramate
- Topamax (Active Comparator)
  Interventions: Drug: topiramate

INTERVENTIONS:
Drug: topiramate — Topiramate (brand name Topamax) is an anticonvulsant (antiepilepsy) drug. IUPAC name 2,3:4,5-Bis-O-(1-methylethylidene)-beta-D-fructopyranose sulfamate

SUMMARY:
* Objective:

  * Compare the bioequivalence of a test topiramate formulation (Torrent Pharmaceuticals Limited) to an equivalent oral dose of the commercially available topiramate (Topamax®, Ortho-McNeil Neurologics, Inc.) in a test population of adult subjects under fed conditions.
* Clinical Design:

  * Studies were Randomized, Two-Way Crossover, Single-Dose,Open-Label in healthy human adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female; similar proportions of each preferred.
* Age: At least 18 - 55 years (inclusive).
* Weight: BMI (Body Mass Index) 19 kg/m2 - 30 kg/m2 (inclusive).
* Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory tests, all obtained within four (4) weeks prior to study start. The subject may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:

  1. Laboratory Tests: Serum pregnancy test (female subjects only), hemoglobin, hematocrit, RBC, WBC, platelet count, differential count, serum electrolytes (Na, K, Cl), fasting blood glucose, BUN, bilirubin, creatinine, AST, ALT, LD, alkaline phosphatase, urinalysis, drugs of abuse, HIV, Hepatitis B, and Hepatitis C will be done for screening purposes.Laboratory values which are greater than 20% of the normal range will not qualify unless specifically accepted by a physician who is an investigator or sub-investigator for the clinical trial. Results of a serum pregnancy test (female subjects only), HIV, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study.
  2. Electrocardiogram A 12-lead electrocardiogram (ECG) will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
* Subjects must read and sign the Consent Form.

Exclusion Criteria:

* Subjects not complying with the above inclusion criteria must be excluded from the study.
* In addition, any one (1) of the conditions listed below will exclude a subject from the study:

  1. History of treatment for alcoholism, substance abuse, or drug abuse within the past 24 months.
  2. History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
  3. History of GERD (gastroesophageal reflux disease), malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
  4. History of treatment for asthma within the past five (5) years.
  5. History of predisposition to renal calculi.
  6. History of surgery within the past eight (8) weeks.
  7. History of application of tattoo(s) within the past 30 days.
  8. History of body piercing(s) within the past 30 days.
  9. Females who are pregnant or lactating.
  10. History of hypersensitivity to topiramate or any anticonvulsant medication.
* Conditions upon screening which might contraindicate or require that caution be used in the administration of topiramate, including:

  1. Sitting systolic blood pressure below 90 mm Hg, or diastolic pressure below 50 mm Hg.
  2. Heart rate less than 50 beats per minute after a 5-minute rest in a seated position.
* Inability to read and/or sign the consent form.
* Treatment with any other investigational drug during the 30 days prior to the initial dosing for this study.
* Subjects who have donated blood within 30 days prior to the initial dosing for this study.
* Subjects who smoke more than 10 cigarettes per day.
* Subjects who do not tolerate venipuncture.
* Subjects who have difficulty fasting or consuming standardized meals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Torrent's Topiramate First, Then Topamax: For period one - on the morning of Day 1 subjects received two tablets of the test formulation, Torrent's Topiramate 25 mg.
  Followed by a 21 day washout period.
  For period two - on the morning of Day 1 subjects received two tablets of the reference formulation, Topamax 25 mg.
- Topamax First, Then Torrent's Topiramate: For period one - on the morning of Day 1 subjects received two tablets of the reference formulation, Topamax 25 mg.
  Followed by a 21 day washout period.
  For period two - on the morning of Day 1 subjects received two tablets of the test formulation, Torrent's Topiramate 25 mg.
Period: Period 1 - First Intervention - 5 Days
Arm/Group | Torrent's Topiramate First, Then Topamax | Topamax First, Then Torrent's Topiramate
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2 - Washout Period - 21 Days
Arm/Group | Torrent's Topiramate First, Then Topamax | Topamax First, Then Torrent's Topiramate
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 3 - Second Intervent - 5 Days
Arm/Group | Torrent's Topiramate First, Then Topamax | Topamax First, Then Torrent's Topiramate
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Torrent's Topiramate: tablet containing 25 mg of topiramate (Torrent Pharmaceuticals Limited.Administered at Hour 0 on Day 1 of each test period.
- Topamax: tablet containing 25 mg of topiramate (Topamax®, Ortho-McNeil Neurologics, Inc.), to be administered at Hour 0 on Day 1 of each test period.
- Total: Total of all reporting groups
Arm/Group | Torrent's Topiramate | Topamax | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.8) | 32.4 (10.8) | 32.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after drug administration.
Population: Pharmacokinetic analyses are based on 18 out of 18 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng / ml
Units Other Than Participants: blood samples
Arm/Group | Torrent's Topiramate | Topamax
Number analyzed (Participants) | 18 | 18
Number analyzed (blood samples) | 396 | 396
ng / ml | 270.31 (100.30) | 248.46 (85.69)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t)
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses are based on 18 out of 18 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng h / ml
Units Other Than Participants: blood samples
Arm/Group | Torrent's Topiramate | Topamax
Number analyzed (Participants) | 18 | 18
Number analyzed (blood samples) | 396 | 396
ng h / ml | 13762.05 (4003.49) | 13152.04 (3478.45)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses are based on 18 out of 18 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng h / ml
Units Other Than Participants: blood samples
Arm/Group | Torrent's Topiramate | Topamax
Number analyzed (Participants) | 18 | 18
Number analyzed (blood samples) | 396 | 396
ng h / ml | 19689.88 (5889.87) | 18088.71 (4390.57)

ADVERSE EVENTS:
Time Frame: 1 month
Description: 18 out of 18 enrolled subjects completed this study.
Arm/Group | Torrent's Topiramate | Topamax
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Torrent's Topiramate (N=18) | Topamax (N=18)
Dizziness (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Intermediate Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hematoma (Right Arm) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other